CLINICAL TRIAL: NCT01938599
Title: A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study Comparing AM001 Cream to Vehicle in the Treatment of Plaque Psoriasis
Brief Title: Study Comparing AM001 Cream to Vehicle in the Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AmDerma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AD-AM001-001
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Plaque Psoriasis; Skin Diseases, Papulosquamous; Skin Diseases
Keywords: Plaque Psoriasis
MeSH Terms: conditions — Skin Diseases, Papulosquamous; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AM001 (Experimental): AM001 Cream, 7.5%. 2x daily for 12 weeks.
  Interventions: Drug: AM001 Cream, 7.5%
- Vehicle (Placebo Comparator): Placebo of AM001 Cream. 2x daily for 12 weeks.
  Interventions: Drug: Placebo of AM001 Cream

INTERVENTIONS:
Drug: AM001 Cream, 7.5% — Cream, 2x daily for 12 weeks
  Arms: AM001
Drug: Placebo of AM001 Cream — Cream, 2x daily for 12 weeks
  Arms: Vehicle

SUMMARY:
To compare the safety and efficacy profile of AM001 Cream and its vehicle in the treatment of plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide Institutional Review Board (IRB) approved written informed consent.
2. Subjects must be male or female, at least 18 years of age.
3. Subjects with a definite diagnosis of plaque psoriasis that is clinically active (for at least 3 months), involving at least 3% and up to 20% of the body surface area (not including the scalp, face, hands, feet, and intertriginous areas).
4. Subjects with an Investigator's Global Assessment (IGA) of disease severity of at least moderate severity (score ≥ 3) as an overall assessment.
5. Subjects with a minimum plaque elevation of at least moderate severity (PASI grade ≥ 3) at the target lesion site.
6. If females of childbearing potential, the subject must have a negative urine pregnancy test, and must have been using an acceptable form of birth control for at least two months prior to Screening and are willing to continue birth control throughout the study.
7. Subjects must be willing and able to understand and comply with the requirements of the study, apply the study medication as instructed, return for the required treatment period visits, comply with therapy prohibitions, and be able to complete the study.
8. Subjects must be in good health, as confirmed by medical history and physical exam, and free from any clinically significant disease/condition, other than plaque psoriasis, that might interfere with the study evaluations.
9. Subjects must be willing to limit sun exposure overall. Subjects are prohibited from sunbathing or intentional tanning or intense sun exposure including the use of tanning booths/lights or other artificial UV light sources throughout the study.

Exclusion Criteria:

1. Female subjects who are pregnant, nursing, or planning a pregnancy within the study participation period.
2. Subjects who have a current diagnosis of guttate, pustular, inverse, exfoliative, or erythrodermic psoriasis.
3. Subjects who have a history of psoriasis unresponsive to topical treatments.
4. Subjects who have a history of a disorder that may interfere with the evaluation of plaque psoriasis (e.g., atopic dermatitis, contact dermatitis, tinea corporis, cutaneous lymphoma, etc.).
5. Presence of pigmentation, extensive scarring, or pigmented lesions in the treatment areas, which could interfere with the rating of efficacy parameters.
6. Subjects with unstable medical disorders, life-threatening disease, or current malignancies.
7. Subjects with clinically significant ECG or laboratory abnormalities at Screening (as determined by the Investigator).
8. Subjects who are immunosuppressed.
9. Subjects who have a history of allergy or a known hypersensitivity to any component of the study medication.
10. Subjects who have been treated with any systemic steroids within the 4 weeks prior to the study entry.
11. Subjects who have been treated with systemic or photo antipsoriatic therapies/drugs within 4 weeks prior to study entry including methotrexate, cyclosporine, acitretin and other oral retinoids, broadband or narrowband UVB, PUVA, home or professional tanning lights or other nonprescription UV light sources, photodynamic therapy (PDT), lasers, mycophenalate mofetil (MMF), thioguanine, hydroxyurea, sirolimus, azathioprine, 6-mercaptopurine (6-MP), or etanercept.
12. Subjects who have been treated with biologic therapy other than etanercept within 8 weeks prior to study entry. Vaccines will not be considered an exclusionary biologic treatment.
13. Subjects who have been treated with any topical anti-psoriatic (e.g., salicylic acid, anthralin, tar, etc.,) any topical corticosteroid medications, topical retinoids (e.g., tazarotene, tretinoin), topical Vitamin D analogs (e.g., calcipotriene), topical immunosuppressants (e.g., tacrolimus, pimecrolimus) within 2 weeks prior to study entry.
14. Subjects who have been treated with lithium, antimalarial agents, or quinidine within the 4 weeks prior to study entry.
15. Subjects who have received radiation therapy and/or anti-neoplastic agents, or taken any immunosuppressant medication within 3 months prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment of Disease Severity (IGA) | Week 12
  An overall assessment of disease severity will be performed at each study visit.

SECONDARY OUTCOMES:
Target Lesion Psoriasis Area Severity Index (PASI) | 12 Weeks
  Erythema, Scaling and Plaque Elevation of the target lesion will be scored at baseline and at each subsequent study visit.
Body Surface Area (BSA) | 12 Weeks
  The % BSA of all treatable psoriatic lesions and regions will be recorded at baseline and at week 12.
Target Lesion Area | 12 Weeks
  The target lesion area will be measured at baseline and each-post-baseline visit.
Dermatology Life Quality Index (DLQI) | 12 Weeks
  Measured at baseline and week 12.
Pharmacokinetics | 2 Weeks
  Systemic absorption will be determined in a subgroup.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - International Dermatology Research, Inc., Miami, Florida
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Association, Albuquerque, New Mexico
  - Dermatology Consulting Services, High Point, North Carolina
  - J & S Studies, College Station, Texas